CLINICAL TRIAL: NCT05576220
Title: Remote Temperature Monitoring of Adult Subjects Undergoing Outpatient Stem Cell Transplant or CAR-T Cell Therapy at Risk for Developing Infections and/or Cytokine Release Syndrome
Brief Title: Remote Temperature Monitoring of Adult Subjects Undergoing Outpatient Stem Cell Transplant or CAR-T Cell Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IDION Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IDN001
Record Dates: First submitted 2022-10-02; First posted 2022-10-12 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Febrile Neutropenia
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention group (Experimental): Subjects being treated for a cancer diagnosis with a plan for outpatient transplant or CAR-T therapy
  Interventions: Device: IDION iTempShield
- Control Group (No Intervention): Retrospective data from the control group comprised of 105 patients directly preceding the intervention group who are underwent stem cell transplant or CAR-T therapy. Such control group information will be obtained via a research data request. Only de-identified data will be obtained for these subjects.

INTERVENTIONS:
Device: IDION iTempShield — Subject is being treated for a cancer diagnosis with a plan for outpatient transplant or CAR-T therapy
  Arms: Intervention group

SUMMARY:
IDION is currently seeking FDA approval for this device- the IDION iTempShield. It is a skin-safe, FDA complaint and non-invasive device that can read and monitor skin temperature. Having continuous temperature monitoring using the IDION iTempShield may provide early detection of a fever for patients with febrile neutropenia. Febrile neutropenic fever is common in patients receiving chemotherapy and can often indicate infection. The main potential benefit potenially experienced from participating in this study would be the early detection of fever.

There is a potential benefit that infection will be detected earlier in subjects wearing the IDION iTempShield.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the remote patient temperature monitoring service of the Idion Shield system in patients undergoing outpatient stem cell transplantation or CAR-T therapy who are at risk for developing infections and/or cytokine release syndrome. Febrile neutropenia remains a significant complication of treatment and often it is the first and sometimes the only sign or symptom of infection in this vulnerable patient population.

CAR-T patients are at risk for not only febrile neutropenia but also cytokine release syndrome (CRS), a systemic inflammatory response that can lead to hypoxia and shock. Fever is typically the first sign and hallmark of this potentially life-threatening condition. Routine measurement of body temperature is an important aspect of monitoring for signs of infection in patients receiving chemotherapy and for CRS in CAR-T patients.The current of standard of care for patients is to take their oral temperature when they feel ill and directing them to call their physician when their oral temperature reading is above 100.4. Having continuous temperature monitoring using the IDION iTempShield may provide early detection and intervention while reducing hospitalization rates, improving outcomes, and preventing death. With an increase in technological advancements and telemedicine, remote monitoring has shown to reduce health costs while providing closer follow-up for patients. The study will also analyze the potential reimbursement through Medicare to show the cost-benefit for remote monitoring utilizing the IDION iTempShield.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is being treated for a cancer diagnosis with a plan for outpatient transplant or CAR-T therapy
2. Subject is ≥ 18 years or older.
3. Subject is being treated or coming to the infusion center for clinical follow up every 2 weeks.
4. Subject has an iOS or Android phone.
5. Subject is willing to install the Idion app on his/her phone.
6. Subject self identifies as proficient in smart phone use.
7. Subject is willing to allow Idion to send text reminders to take temperature or complete surveys.
8. Subject is willing to configure the phone to ensure these notifications are delivered, even when phone is in a "no notification" mode.
9. Subject or subject caretaker is able and willing to complete subject surveys.
10. Subject is willing and able to provide written informed consent in English or Spanish.
11. Subject is willing and able to comply with all study procedures, requirements, assessments, visits, and complete questionnaires.

Exclusion Criteria:

1. Non-English or Spanish speakers
2. Unable to provide informed consent
3. Subjects with known adhesive allergy for silicon adhesives
4. Subjects with history of Medical Adhesive-Related Skin Injury (MARSI)
5. Subjects with no available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the IDION Shield remote subject temperature monitoring service. | 6 Months
  The ability of the Idion System to transmit alerts if there is a temperature excursion sustained for at least 15 minutes above the alert protocol. There is a full data set time correlated with temp data in, battery voltage status and alerts that have been sent by Idion. The data will be mined and compared with the number of alerts and the timing of those alerts in the database.There will be times when the mobile device is offline due to mobile device battery exhaustion or distance traveled away from the device (left mobile at home) and these alerts will be missed.
To evaluate the IDION Shield remote subject temperature monitoring service. | 6 Months
  The accuracy of the Idion iTempShield as validated by subject taking their temperature manually with the thermometer, to be captured in the subject app. This data is transmitted to the clinician application, and this will demonstrate subject use and shield interoperability.
To evaluate the IDION Shield remote subject temperature monitoring service. | 6 Months
  The ability of the Idion iTempShield to be paired with the subject's phone. This data will be subjective data.This endpoint will be calculated as the number of successful pairings (i.e., where pairing was confirmed by Idion System) divided by the total number of pairing attempts. The point estimate of the successful pairings along with a 90% confidence interval will be presented.
To evaluate the IDION Shield remote subject temperature monitoring service. | 6 Months
  Test alert protocol with clinicians pre-pilot to simulate an alert event. Testing will entail inputting a manual temperature of over 100.4 into the patient app. If the clinician receives a phone call, text, or email alerting them that there has been a temperature event, this test will be deemed successful. If this is not functioning properly the software will be adjusted and a new test will be performed. If this cannot be done, then the Pilot will be paused until corrected.
To evaluate the IDION Shield remote subject temperature monitoring service. | 6 Months
  The incidence of Idion iTempShield-alerted temperature events in the overnight hours (9pm-6am and 12am-6am). Analyze temperature trends and clinical course at 3 hours pre and post alert and 6 hours pre and post alert. This is not the normal course of treatment for these subjects. This data set is an attempt to uncover temperature trends that may change the course of treatment for cancer patients.

SECONDARY OUTCOMES:
To evaluate the clinical course of subjects with elevated temperatures | 6 Months
  Review the treatment course of all subjects participating in the study to determine if any subjects received treatment as a response to the temperature alert and what percentage of these subjects went to the hospital. Review the treatment course for those who were admitted from admission to discharge of subjects who were admitted due to a temperature excursion. This data will need to be pulled from two asynchronous source the EMR and the Clinician Application. The information that is being compared is outpatient or admission to hospital.
To evaluate the clinical course of subjects with elevated temperatures | 6 Months
  Compare the level of care for chemotherapy patients admitted to the hospital wearing the iTempShield versus those not wearing the iTempShield. Level of care will focus specifically on whether or not patients were admitted to the ICU upon admission to the hospital and if they were being treated for sepsis. The "control group" will comprise of up to 105 patients who are undergoing stem cell transplant or CAR-T therapy. Subjects in the control group will be identified via retrospective chart review and data collected on these subjects will be done in a de-identified manor. The "control group" will comprise of 105 patients directly preceding the intervention group who are undergoing stem cell transplant or CAR- T therapy. The control group of subjects will be compared to those in the intervention group. The level of care will focus specifically on whether subjects were admitted to the ICU upon admission to the hospital and if they were being treated for sepsis.
To assess subject and clinician satisfaction and compliance with the remote subject temperature monitoring service. | 6 Months
  Subject and clinician satisfaction (based on surveys).
To assess subject and clinician satisfaction and compliance with the remote subject temperature monitoring service. | 30 days
  Subject and clinician adherence to the protocol; reason for non-adherence, number of subjects who comply and wear the Shield for the entire 30 days.

OTHER OUTCOMES:
To analyze reimbursement for remote subject management. | 6 Months
  Amount of Medicare reimbursement potential. The clinician app will automatically enroll the patient into a CMS approved reimbursement, and we also track their insurance (private and Medicare) in the application. This information is to determine what potential reimbursements could be.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No